CLINICAL TRIAL: NCT06791460
Title: Pegylated Liposomal Doxorubicin Plus Adebrelimab With or Without Mirabegron in Relapsed Ovarian Cancer: a Randomized, Controlled, Open-label Trial
Brief Title: Pegylated Liposomal Doxorubicin Plus Adebrelimab With or Without Mirabegron in Relapsed Ovarian Cancer
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Obstetrics & Gynecology Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Xin Wu, Deputy Chief of Gynecologic Oncology, Obstetrics & Gynecology Hospital of Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUOBGY-2024-154
Record Dates: First submitted 2025-01-17; First posted 2025-01-24 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-01

CONDITIONS: Ovarian Cancer Recurrent
MeSH Terms: interventions — liposomal doxorubicin; mirabegron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pegylated liposomal doxorubicin plus adebrelimab with mirabegron (Experimental)
  Interventions: Drug: Pegylated liposomal doxorubicin plus adebrelimab with mirabegron
- Pegylated liposomal doxorubicin plus adebrelimab (Active Comparator)
  Interventions: Drug: Pegylated liposomal doxorubicin plus adebrelimab

INTERVENTIONS:
Drug: Pegylated liposomal doxorubicin plus adebrelimab with mirabegron — Participants receive pegylated liposomal doxorubicin at a dose of 20mg/m2 plus adebrelimab at a dose of 20 mg/kg via intravenous (IV) infusion plus on Day 1 of each 21-day cycle orally with daily mirabegron until intolerance or disease progression.
  Arms: Pegylated liposomal doxorubicin plus adebrelimab with mirabegron
Drug: Pegylated liposomal doxorubicin plus adebrelimab — Participants receive pegylated liposomal doxorubicin at a dose of 20mg/m2 plus adebrelimab at a dose of 20 mg/kg via intravenous (IV) infusion plus on Day 1 of each 21-day cycle until intolerance or disease progression.
  Arms: Pegylated liposomal doxorubicin plus adebrelimab

SUMMARY:
The goal of this clinical trial is to learn if drug regimen pegylated liposomal doxorubicin and adebrelimab with or without mirabegron works to treat relapsed ovarian cancer in adults. It will also learn about the safety of drug regimen pegylated liposomal doxorubicin and adebrelimab with or without mirabegron. The main questions it aims to answer are:

Does drug pegylated liposomal doxorubicin and adebrelimab with or without mirabegron reduce tumor volume? What medical problems do participants have when taking drug pegylated liposomal doxorubicin and adebrelimab with or without mirabegron?

Researchers will compare drug regimen pegylated liposomal doxorubicin and adebrelimab with mirabegron to a drug regimen pegylated liposomal doxorubicin and adebrelimab without mirabegron to see which drug regimen works better to treat relapsed ovarian cancer.

Participants will:

Take drug pegylated liposomal doxorubicin and adebrelimab every 21 days with or without everyday mirabegron Visit the clinic once every 2 months for checkups and tests Keep a diary of their symptoms

ELIGIBILITY:
Inclusion Criteria:

* Has provided documented informed consent for the study.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Has histologically confirmed epithelial ovarian, fallopian tube, or primary peritoneal carcinoma.
* Has received a front line platinum-based regimen (administered via either intravenous or intraperitoneal route) per local standard of care or treatment guideline following the primary or interval debulking surgery with documented disease recurrence (note: Maintenance treatment following the front line treatment is permitted and counted together as part of the front line treatment).
* Has a platinum-free interval (PFI) of < 12 months if the last regimen received is a platinum-based, or a treatment-free interval (TFI) of < 12 months if the last regimen received is a non-platinum-based.
* Has measurable disease at baseline based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
* Has a life expectancy of ≥12 weeks.
* Has provided a tumor tissue sample either collected from prior cytoreductive surgery or fresh newly obtained tumor tissue at screening.
* Has adequate organ function.
* Has not recovered from AEs to ≤ Grade 1 or prior treatment level due to a previously administered agent.

Exclusion Criteria:

* Has nonepithelial cancers, borderline tumors, mucinous, seromucinous that is predominantly mucinous, malignant Brenner's tumor and undifferentiated carcinoma.
* Has received prior therapy with an anti-programmed cell death (PD)-1, anti-PD-L1, anti-PD-L2 agent or with an agent directed to another co-inhibitory T-cell receptor (e.g. cytotoxic T-lymphocyte-associated antigen-4 [CTLA-4], tumor necrosis factor receptors OX-40 or CD137) or has participated in prior adebrelimab studies.
* Has received prior systemic anticancer therapy including radiation therapy or maintenance therapy within 4 weeks before randomization.
* Has severe hypersensitivity (≥Grade 3) or uncontrolled hypertension to pegylated liposomal doxorubicin, adebrelimab, mirabegron and any of their excipients.
* Has undergone major surgery within 3 weeks before randomization or has complications/sequelae that have not yet recovered.
* Has a known additional malignancy that progressed or required active treatment within the last 5 years.
* Is pregnant or breastfeeding.
* Has a history of allogenic tissue/solid organ transplant.
* Has a history of thrombotic disorders, hemorrhage, hemoptysis, or active gastrointestinal bleeding within 6 months before randomization.
* Has a history of active autoimmune disease.
* Has an active infection requiring systemic therapy.
* Has a history of human immunodeficiency virus (HIV) infection.
* Has a history of Hepatitis B or C virus infection.
* Has a history or current evidence of any condition, therapy, laboratory abnormality, or other circumstance that might confound the results of the study.
* Has a known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 296 (Estimated)
Dates: Start 2025-03-18 (Estimated); Primary Completion 2028-02-14 (Estimated); Study Completion 2030-02-14 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Month 6
  Objective Response Rate (ORR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) by Blinded Independent Central Review (BICR). ORR was defined as the percentage of participants who had a Complete Response (Disappearance of all target lesions) or a Partial Response (≥30% decrease in the sum of the longest diameter of target lesions) using RECIST 1.1 based on BICR.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) at 6 Months | Month 6
  PFS was defined as the time from first dose of study treatment to the first documented progressive disease (PD) per RECIST 1.1 based on BICR, or death due to any cause, whichever occurred first. Per RECIST 1.1 PD was defined as ≥20% increase in SOD of target lesions and an absolute SOD increase of ≥5 mm.
  The appearance of ≥1 new lesion is also PD. PFS at 6 months is defined as the percentage of patient who was progression free at 6 months from the randomization.
Overall Survival (OS) at 6 Months | Month 6
  OS at 6 months is defined as the percentage of patients who are alive at 6 months from the randomization.
Progression Free Survival (PFS) at 12 Months | Month 12
  PFS was defined as the time from first dose of study treatment to the first documented progressive disease (PD) per RECIST 1.1 based on BICR, or death due to any cause, whichever occurred first. Per RECIST 1.1 PD was defined as ≥20% increase in SOD of target lesions and an absolute SOD increase of ≥5 mm.
  The appearance of ≥1 new lesion is also PD. PFS at 12 months is defined as the percentage of patient who was progression free at 12 months from the randomization.
Overall Survival (OS) at 12 Months | Month 12
  OS at 12 months is defined as the percentage of patients who are alive at 12 months from the randomization.
Incidence of grade 3-4 Adverse Events (AEs) | up to 1 month after the end of treatment
  Incidence of grade 3-4 AEs, according to CTCAE, version 5.0

OTHER OUTCOMES:
Exploratory outcome: biomarkers testing and efficacy of anti-tumor immunity | Baseline and 6 months from the randomization
  Biomarker testing for PD-L1 expression in exploratory analysis.
Exploratory outcome: biomarkers testing and efficacy of anti-tumor immunity | Baseline and 6 months from the randomization
  Biomarker testing for BMI (weight and height will be combined to report BMI in kg/m^2) in exploratory analysis.
Exploratory outcome: biomarkers testing and efficacy of anti-tumor immunity | Baseline and 6 months from the randomization
  Biomarker testing for tumor microenvironment (including density and state of CD8+ T cells density and other immune cells) in exploratory analysis.
Exploratory outcome: biomarkers testing and efficacy of anti-tumor immunity | Baseline and 6 months from the randomization
  Biomarker testing for circulating anti-tumor immunity (including density and state of CD8+ T cells density and other immune cells) in exploratory analysis.
Exploratory outcome: biomarkers testing and efficacy of anti-tumor immunity | Baseline and 6 months from the randomization
  Biomarker testing for transcriptome in exploratory analysis.
Exploratory outcome: biomarkers testing and efficacy of anti-tumor immunity | Baseline and 6 months from the randomization
  Biomarker testing for genome in exploratory analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Obstetrics and Gynecology Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No